CLINICAL TRIAL: NCT06430762
Title: Identification of Therapeutic Exposures and Risk Factors Associated With Medication-Related Osteonecrosis of the Jaw
Brief Title: Therapeutic Exposures and Risk Factors in MRONJ
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Principal Investigator, Marmara University
Other Study IDs: CIBON-MAR-A.1
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Medication-Related Osteonecrosis of Jaw

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focuses on patients who have developed a condition called medication-related osteonecrosis of the jaw (MRONJ), which can occur after using certain medications. The purpose is to closely monitor these patients over time to better understand how they are diagnosed, treated, and followed up. By doing this, researchers hope to uncover how different factors such as a patient's background, lifestyle, and other health conditions might influence their recovery and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Male or female individuals
* Individuals who apply to the Marmara University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery due to medication-related osteonecrosis of jaw during the study period
* Individuals or their legal representatives who have given written consent to participate in the study

Exclusion Criteria:

* Non-drug-related osteonecrosis/osteomyelitis
* Osteoradionecrosis
* Metastasis to the oral region
* Individuals who have not given written consent to participate in the study
* Individuals under the age of 18

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this research comprises individuals aged 18 and over, both male and female, who present with medication-related osteonecrosis of the jaw (MRONJ) at the Oral and Maxillofacial Surgery Clinic of Marmara University Faculty of Dentistry. The study excludes individuals with non-drug-related osteonecrosis or osteomyelitis, osteoradionecrosis, those with metastasis to the oral region, individuals who have not provided consent, and those under the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
Change in Karnofsky Performance Status | 24 months
  This outcome measures the overall health status and activity levels of patients with MRONJ using the Karnofsky Performance Scale (KPS). KPS rates patients on a scale from 0 to 100, where higher scores indicate greater independence and lower morbidity risk, while lower scores reflect dependency and the need for substantial medical intervention. The scale's aim is to quantify the extent to which patients can perform everyday life activities without assistance. At baseline (T0), 3 months (T1), 6 months (T2), 12 months (T3), 18 and 24 months (T4, if required), the questionnaire will be taken.
Change in Oral Health-related Quality of Life | 24 months
  A scale of 1 to 5 will be used to rate each of the 14 questions about how dental health affects quality of life (minimum score of 0, maximum score of 70). Higher ratings reflect a greater influence of the patient's dental health on their quality of life (higher scores, worse outcomes). At baseline (T0), 3 months (T1), 6 months (T2), 12 months (T3), 18 and 24 months (T4, if required), the questionnaire will be taken.
Change in staging of MRONJ | 24 months
  Staging of the lesion in the mouth will be according to the definition of the American Association of Oral and Maxillofacial Surgeons (Ruggiero et al. 2022). Clinical examination will be performed at baseline (T0), 3 months (T1), 6 months (T2), 12 months (T3), 18 and 24 months (T4, if necessary).
Biochemical Markers Related to Bone Metabolism and Inflammatory Response | Baseline
  Various biochemical markers indicative of bone metabolism and inflammatory response in patients with medication-related osteonecrosis of the jaw (MRONJ) will be evaluated. The markers include serum calcium, ionized calcium, parathyroid hormone (PTH), alkaline phosphatase, osteocalcin, C-telopeptide (CTX), Vitamin D3, C-reactive protein (CRP), and leukocyte count. Blood samples collected at baseline will be analyzed.
Change in the Assessment of Radiographic Changes Using the Composite Radiographic Index | 24 months
  This outcome involves utilizing the Composite Radiographic Index to track and characterize the progression of lesions in patients with medication-related osteonecrosis of the jaw. This index evaluates:
  * Location of the lesion: Maxilla anterior, Maxilla posterior, Mandible anterior, Mandibular posterior.
  * Lyric changes: Scored as 0 (None), 1 (Localized), 2 (Widespread).
  * Sclerosis: Scored as 0 (None), 1 (Localized), 2 (Widespread).
  * Periosteal bone formation: Scored as 0 (None), 1 (Localized), 2 (Widespread).
  * Sequestration: Scored as 0 (None), 1 (Localized), 2 (Widespread). Radiographs will be taken at the initial visit to establish a baseline for each patient. Subsequent radiographs will be taken only if clinically indicated to monitor the presence and progression of osteonecrotic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Ferit Bayram, PhD, Study Chair — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruggiero SL, Dodson TB, Aghaloo T, Carlson ER, Ward BB, Kademani D. American Association of Oral and Maxillofacial Surgeons' Position Paper on Medication-Related Osteonecrosis of the Jaws-2022 Update. J Oral Maxillofac Surg. 2022 May;80(5):920-943. doi: 10.1016/j.joms.2022.02.008. Epub 2022 Feb 21. PMID 35300956
- [Background] Friendlander AH, Ettinger RL. Karnofsky performance status scale. Spec Care Dentist. 2009 Jul-Aug;29(4):147-8. doi: 10.1111/j.1754-4505.2009.00088.x. No abstract available. PMID 19573040
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805